CLINICAL TRIAL: NCT07013890
Title: Effectiveness and Safety of an Association of Phycocyanin and Palmitoylethanolamide in Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: A Prospective Observational Multicentric Study
Brief Title: Efficacy of Phycocyanin and Palmitoylethanolamide for the Treatment of Chronic Prostatitis Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Urologica Molinette - Città della Saliute e della Scienza (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other)
Responsible Party: Principal Investigator, Mattia Sibona, Urologist, MD, Clinica Urologica Molinette - Città della Saliute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CET n. 530/2021
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-01

CONDITIONS: Chronic Prostatitis (CP); Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Chronic Prostatitis/ Pelvic Pain Syndrome
Keywords: Chronic prostatitis; chronic pelvic pain syndrome; LUTS; pain; phycocyanin; palmitoylethanolamide; FICOXPEA®; phytotherapy
MeSH Terms: conditions — Prostatitis; Pain | interventions — palmidrol; Selenium

STUDY DESIGN:
Intervention Model Description: prospective, observational, multicentric, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FICOXPEA® (Experimental): FICOXPEA® is a phytoterapic compound made of:
  * phycocyanin (spirulina platensis extract) 250 mg
  * palmitoylethanolamide 200 mg
  * L-selenometionine 11 mg
    1. capsule containing all these compounds is administered every day for 30 days
  Interventions: Drug: FICOXPEA® is an oral combination of Phycocyanin, Palmitoylethanolamide and selenium

INTERVENTIONS:
Drug: FICOXPEA® is an oral combination of Phycocyanin, Palmitoylethanolamide and selenium — FICOXPEA® is a phytoterapic compound made of:
  * phycocyanin (spirulina platensis extract) 250 mg
  * palmitoylethanolamide 200 mg
  * L-selenometionine 11 mg

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is a bothering condition characterized by pain localized to the pelvic, perineal and/or genital area and lower urinary tract symptoms (LUTS). Phytotherapy, which involves the combination of two or more active compounds, can be used to treat this challenging condition.

The aim of this study was to investigate the role of an association of phycocyanin (PC) and palmitoylethanolamide (PEA) and selenium (FICOXPEA®) in male patients affected by CP/CPPS.

The main questions the present study aims to answer are:

* Does FICOXPEA® enhance quality of life of CPP/CPPS patients?
* Does it help reducing pain symptoms of CPP/CPPS patients?

Researchers will investigate whether FICOXPEA® works to treat CPP/CPPS symptoms, so its efficacy, but also its tolerability and adherence to therapy.

Participants will:

* Take FICOXPEA® once a day for 30 days;
* Visit the clinic for follow-up visits at 1 and 3 months;
* Answer validated questionnaires and declare potential adverse events at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* adult male patients (aged >18 years)
* clinical affection by CP/CPPS with symptoms that persisted for ≥ 3 months;
* PSA values of 4 to 10 ng/ml (at least 2 determinations)
* patients must have completed diagnostic work-up, such as multiparametric prostate MRI (evidence level 1a according to EAU guidelines) with or without subsequent prostate biopsy (according to the diagnostic flow-chart depicted by EAU international guidelines).

Exclusion Criteria:

* patients with previous diagnosis of prostate cancer
* patients who underwent previous low urinary tract surgery
* patients who underwent previous intravescical chemotherapy
* patients with acute bacterial prostatitis
* diagnostic work-up for prostate cancer not completed
* patients having antibiotic therapy or specific chronic prostatis treatment (phytotherapy included) or benign prostatic iperplasia treatment (e.g. alpha litics) at the time of the recruitment or finished less than a month before

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients (with a prostate)
Enrollment: 48 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Statistically significant change of CPSI total score compared to baseline | 1 month and 3 months
  Improvement of CP symptoms

SECONDARY OUTCOMES:
Statistically significant change of CPSI pain domain score compared to baseline | 1 month and 3 months
  improvement of CP pain symptoms
Statistically significant change of CPSI QoL domain score compared to baseline | 1 month and 3 months
  Improvement of CP QoL
Statistically significant change of total PSA | 1 month and 3 months
  Decrease of chronic altered PSA values
n° of any adverse events | 1 month and 3 months
  number and type, so safety analysis

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Molinette Hospital, Torino, Torino
  - Dipartimento di Chirurgia Università di Catania, Catania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagenlehner FM, Schneider H, Ludwig M, Schnitker J, Brahler E, Weidner W. A pollen extract (Cernilton) in patients with inflammatory chronic prostatitis-chronic pelvic pain syndrome: a multicentre, randomised, prospective, double-blind, placebo-controlled phase 3 study. Eur Urol. 2009 Sep;56(3):544-51. doi: 10.1016/j.eururo.2009.05.046. Epub 2009 Jun 3. PMID 19524353
- [Background] Litwin MS, McNaughton-Collins M, Fowler FJ Jr, Nickel JC, Calhoun EA, Pontari MA, Alexander RB, Farrar JT, O'Leary MP. The National Institutes of Health chronic prostatitis symptom index: development and validation of a new outcome measure. Chronic Prostatitis Collaborative Research Network. J Urol. 1999 Aug;162(2):369-75. doi: 10.1016/s0022-5347(05)68562-x. PMID 10411041
- [Background] Sibona M, Destefanis P, Agnello M, Lillaz B, Giuliano M, Cai T, Gontero P. The association of Boswellia resin extract and propolis derived polyphenols can improve quality of life in patients affected by prostatitis-like symptoms. Arch Ital Urol Androl. 2020 Jan 14;91(4):251-255. doi: 10.4081/aiua.2019.4.251. PMID 31937091
- [Background] Cai T, Luciani LG, Caola I, Mondaini N, Malossini G, Lanzafame P, Mazzoli S, Bartoletti R. Effects of pollen extract in association with vitamins (DEPROX 500(R)) for pain relief in patients affected by chronic prostatitis/chronic pelvic pain syndrome: results from a pilot study. Urologia. 2013 Apr 24;80 Suppl 22:5-10. doi: 10.5301/RU.2013.10597. Epub 2013 Jan 16. PMID 23334883